CLINICAL TRIAL: NCT00436774
Title: Cross-Sectional Evaluation of Outcome Following Extra-Cranial Germ Cell Tumors Treated According to UKCCSG GC 7901 (GC I) and GC 8901 (GC II) Protocols
Brief Title: Treatment Outcome and Quality of Life in Patients With Pediatric Extra-Cranial Germ Cell Tumors Previously Treated on Clinical Trial CCLG-GC-1979-01 or CCLG-GC-1989-01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CCLG-GC-2006-06; CDR0000531140 (Registry Identifier: PDQ (Physician Data Query)); EU-20642
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-06

CONDITIONS: Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Gastrointestinal Complications; Infertility; Long-term Effects Secondary to Cancer Therapy in Children; Neurotoxicity; Ovarian Cancer; Pulmonary Complications; Sexual Dysfunction; Urinary Complications
Keywords: long-term effects secondary to cancer therapy in children; neurotoxicity; gastrointestinal complications; pulmonary complications; sexual dysfunction; infertility; urinary complications; childhood extragonadal germ cell tumor; childhood malignant ovarian germ cell tumor; childhood malignant testicular germ cell tumor; childhood teratoma
MeSH Terms: conditions — Infertility; Neurotoxicity Syndromes; Ovarian Neoplasms; Sexual Dysfunction, Physiological; Ovarian Germ Cell Cancer; Testicular Neoplasms; Teratoma

INTERVENTIONS:
Procedure: assessment of therapy complications
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Treatment for pediatric extracranial germ cell tumors may cause side effects and secondary cancers later in life. A study that evaluates patients after receiving combination chemotherapy or surgery may help doctors understand the side effects and secondary cancers that occur later in life.

PURPOSE: This study is looking at treatment outcome and quality of life in patients with pediatric extracranial germ cell tumors previously treated on clinical trial CCLG-GC-1979-01 or CCLG-GC-1989-01.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the late effects of treatment and the quality-of-life of patients with germ cell tumors (GCT) previously treated on clinical trial CCLG-GC-1979-01 or CCLG-GC-1989-01.
* Evaluate the late effects of carboplatin, etoposide, and bleomycin in patients treated on clinical trial CCLG-GC-1989-01.
* Determine the toxicity of bleomycin and a combination of either cisplatin and vinblastine, etoposide and cisplatin, or carboplatin and etoposide in patients treated on clinical trial CCLG-GC-1979-01.
* Evaluate tumor-associated/surgical morbidity (bladder, bowel, and lower limb function) in patients with malignant sacrococcygeal tumors treated in these clinical trials.
* Evaluate tumor-associated/surgical morbidity (sexual function/fertility) in patients with malignant gonadal or pelvic GCTs.
* Evaluate tumor-associated/surgical morbidity (respiratory function) in patients with thoracic GCTs.
* Develop a methodology and recommendations for the prospective late evaluation of patients treated on future extracranial GCT clinical trials and those included in this study.
* Inform clinicians about the late effects of treatment of malignant GCTs and advise them on what long-term care these patients require.

OUTLINE: This is a cohort, multicenter study.

Patients complete questionnaires about ototoxicity, bladder and bowel dysfunction, and sexual function and fertility as appropriate. They also complete a health-related quality-of-life questionnaire over 20 minutes.

Treating physicians complete a lower-limb and neurologic dysfunction questionnaire. Data from myelodysplasia, second malignancy, ototoxicity, nephrotoxicity, and pulmonary toxicity assessments are collected from the patient's treating physician.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Previously enrolled in 1 of the following United Kingdom Children's Cancer Study Group (UKCCSG) clinical trials for treatment of extracranial germ cell tumors:

  * CCLG-GC-1989-01
  * CCLG-GC-1979-01

    * Received bleomycin or cisplatin therapy
* At least 5 years since completion of therapy in these clinical trials
* Attending or in contact with a UKCCSG center

  * Patients treated for sacrococcygeal teratomas and discharged from follow-up are eligible
* No recurrent or progressive disease

PATIENT CHARACTERISTICS:

* No patient deemed unsuitable for this study by the treating clinician

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Ototoxicity as measured by audiogram and Health Utilities Index in patients previously treated with cisplatin or carboplatin
Nephrotoxicity as measured by serum magnesium, calcium, and creatinine and glomerular filtration rate in patients previously treated with cisplatin or carboplatin
Myelodysplasia and second malignancies in patients previously treated with etoposide
Pulmonary toxicity as measured by lung function test and respiratory symptom questionnaire in patients previously treated with bleomycin
Bladder and bowel dysfunction, sexual function, and fertility as measured by patient-completed questionnaires and lower limb and neurological dysfunction as measured by clinician-completed questionnaires in patients with pelvic or sacrococcygeal tumors
Quality of life (QOL) as measured by pediatric cancer quality-of-life inventory or Short Form 36 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Adam Glaser, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (13):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (12):
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Great Ormond Street Hospital for Children, London, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales